CLINICAL TRIAL: NCT02438059
Title: SoSu-liv. A Web- and App-based Intervention Study for Health Promotion Among Social and Health Care Workers in Denmark. A Randomized Controlled Trial
Brief Title: SoSu-liv. Mobile Media for Health Promotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Collaborators: PenSam, Denmark (Unknown); Mobile Fitness A/S (Unknown)
Responsible Party: Principal Investigator, Arne Astrup, Professor and Head of Department, University of Copenhagen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: B283
Record Dates: First submitted 2015-04-28; First posted 2015-05-08 (Estimated); Last update posted 2015-05-08 (Estimated); Status verified 2015-05

CONDITIONS: Obesity
Keywords: Inequality in health; workplace health promotion; internet; mobile app; weight loss; intervention; randomized controlled trial
MeSH Terms: conditions — Obesity; Weight Loss | interventions — Amyloid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Access to the SoSu-liv website and app for 38 weeks.
  Interventions: Behavioral: SoSu-liv website and app
- Control (No Intervention): No treatment for 38 weeks.

INTERVENTIONS:
Behavioral: SoSu-liv website and app — A 38 weeks web- and app-based tool for lifestyle changes intervention.
  Arms: Intervention

SUMMARY:
The purpose of this study is to determine whether a web- and app-based tool for health promotion for social and health care workers in Denmark has an effect on body weight (primary outcome), body fat percentage, waist circumference, blood pressure, cholesterol and blood sugar in a 38 week intervention period.

DETAILED DESCRIPTION:
The study was conducted in six municipalities in Denmark from August 2012 - July 2013. In each municipality two to four nursing homes were randomized to either having access to the SoSu-liv tool for 38 weeks, or act as a controls group, that did not receive any treatment. Those municipalities with an even number of nursing homes were randomized in a 1:1 ratio and municipalities with an odd number of nursing homes in a 2:1 ratio. Twelve out of a total of 20 nursing homes were randomized to SoSu-liv, and 8 were randomized to control. The study was divided into two distinct periods. An initial 16 week period including a team competition among the participating nursing homes using the SoSu-liv tool, and a subsequent 22 week period without a competition.

An information meeting was held at each nursing home during work hours, after which each of the employees who was interested in participating completed the consent form. At the baseline examination taking place a few weeks after, the participants underwent a clinical examination (anthropometry, blood pressure and blood sampling values ), and were subsequently introduced to the SoSu-liv tool, altogether taking up 30-45 minutes. After 16 weeks, the clinical examination was repeated, taking about 15 minutes in total. An identical procedure was applied after the total of 38 weeks. The day before each of the 3 clinical examinations, the participants had to spend approximately 10-15 minutes answering an online questionnaire regarding demographic data, health behaviour and general well-being.

The SoSu-liv tool is a web- and app-based tool developed specifically for this particular group of employees. The program has several social features that encourage the users to interact with each other both digitally, physically and orally at the work place. A general overview of the SoSu-life tool is best given by differentiate the tool into four different sections. The social section is an interactive part making it possible to interact with other colleagues using the program. It includes features to send short messages and challenges to other colleagues, join groups and post messages in discussion forums. The functional section is the practical interactive part. It includes features of food registration (calorie counting), exercise registration, establishing new habits, service of text messages-reminders, and the possibility of emailing a question to an expert. The personal section is where the user can track changes in self-reported variables, such as body weight, waist circumference as well as daily amount of smoked cigarettes, and daily general well-being. Other features of the tool include quizzes, health relevant tests, food recipes and food-cinema, as well as a number of information pages on health. Furthermore, the SoSu-liv-tool used a point system where most of the activities performed using the tool gave points to the individual user. During the first 16 weeks, each nursing home formed a team of participants, and each of the users' individual points were added to the teams' total points. For every point collected by the nursery team, a ticket was generated to the team and put in a draw pool. Each month, the team had a chance to win a price by simple draw. The team with the most points after 16 weeks also won a price. In the last 22 week intervention period, points were still collected, but no prices were provided.

ELIGIBILITY:
Inclusion Criteria:

* Employees working under a FOA (a Danish union) agreement in elderly care in Denmark.

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 566 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Body weight | 38 weeks

SECONDARY OUTCOMES:
Body fat percentage (Measured using a bioelectrical impedance) | 38 weeks
  Measured using a bioelectrical impedance
Waist circumference | 38 weeks
Blood pressure | 38 weeks
Cholesterol | 38 weeks
  Capillary whole blood total cholesterol (measured using bedside equipment)
Blood sugar | 38 weeks
  Capillary whole blood glucose (measured using bedside equipment)

CONTACTS AND LOCATIONS:
Overall Officials: Arne Astrup, Professor, Study Director — Head of Department

REFERENCES:
- [Derived] Balk-Moller NC, Poulsen SK, Larsen TM. Effect of a Nine-Month Web- and App-Based Workplace Intervention to Promote Healthy Lifestyle and Weight Loss for Employees in the Social Welfare and Health Care Sector: A Randomized Controlled Trial. J Med Internet Res. 2017 Apr 10;19(4):e108. doi: 10.2196/jmir.6196. PMID 28396303